CLINICAL TRIAL: NCT01686633
Title: A Randomized, Double-Blind, Parallel Group, Multicenter Study of Fluticasone Furoate/Vilanterol 200/25 mcg Inhalation Powder, Fluticasone Furoate/Vilanterol 100/25 mcg Inhalation Powder, and Fluticasone Furoate 100 mcg Inhalation Powder in the Treatment of Persistent Asthma in Adults and Adolescents
Brief Title: An Efficacy and Safety Study of Fluticasone Furoate/Vilanterol (FF/VI) 200/25 Microgram (mcg) , FF/VI 100/25 mcg, and FF 100 mcg in Adults and Adolescents With Persistent Asthma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 116863
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Results first posted 2014-06-06 (Estimated); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Asthma
Keywords: asthma; pharmacogenetics; adult; vilanterol; adolescents; fluticasone furoate
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate; vilanterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm1: Fluticasone Furoate/ Vilanterol 200/25 mcg (Experimental): At Visit 3, eligible subjects for randomization will be stratified according to their baseline FEV1 performed at Visit 3 (<=65% or >65%) and randomized to one of the three treatment arms. Subjects in this arm will receive FF/ VI 200/25 mcg once daily in the evening for 84 days.
  Interventions: Drug: Fluticasone Furoate/ Vilanterol 200/25 mcg
- Arm 2: Fluticasone Furoate/ Vilanterol 100/25 mcg (Experimental): At Visit 3, eligible subjects for randomization will be stratified according to their baseline FEV1 performed at Visit 3 (<=65% or >65%) and randomized to one of the three treatment arms. Subjects in this arm will receive FF/ VI 100/25 mcg once daily in the evening for 84 days
  Interventions: Drug: Fluticasone Furoate/ Vilanterol 100/25 mcg
- Arm 3: Fluticasone Furoate 100 mcg (Experimental): At Visit 3, eligible subjects for randomization will be stratified according to their baseline FEV1 performed at Visit 3 (<=65% or >65%) and randomized to one of the three treatment arms. Subjects in this arm will receive FF 100 mcg once daily in the evening for 84 days
  Interventions: Drug: Fluticasone Furoate 100 mcg

INTERVENTIONS:
Drug: Fluticasone Furoate/ Vilanterol 200/25 mcg — Fluticasone furoate/ vilanterol will be available as 200/25 mcg Novel dry powder inhaler (NDPI) with 30 doses per device and 200/25 mcg per actuation
  Arms: Arm1: Fluticasone Furoate/ Vilanterol 200/25 mcg
Drug: Fluticasone Furoate/ Vilanterol 100/25 mcg — Fluticasone furoate/ vilanterol will be available as 100/25 mcg NDPI with 30 doses per device and 100/25 mcg per actuation
  Arms: Arm 2: Fluticasone Furoate/ Vilanterol 100/25 mcg
Drug: Fluticasone Furoate 100 mcg — Fluticasone furoate will be available as 100 mcg NDPI with 30 doses per device and 100/25 mcg per actuation
  Arms: Arm 3: Fluticasone Furoate 100 mcg

SUMMARY:
This is a Phase III, multicenter, randomized, double-blind, stratified, parallel-group study with three active comparators in subjects with moderate to severe persistent asthma. The study consists of a run-in period of 4 weeks, followed by a treatment period of 12 weeks, and a follow up contact period of one week. The total duration of the study is 17 weeks. 990 subjects will be randomized to one of three treatments (FF/VI Inhalation Powder 200/25 mcg once daily in the evening; FF/VI Inhalation Powder 100/25 mcg once daily in the evening; FF 100 Inhalation Powder once daily in the evening) for 12 weeks. In addition, all subjects will be supplied albuterol/salbutamol inhalation aerosol at Visit 1 to use as needed for acute asthma symptoms throughout the entire study. Subjects will attend four on-treatment visits at Weeks 2, 4, 8, and 12 (Visits 4 through 7).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must give their signed and dated (written) informed consent to participate. Written informed consent must be obtained if a subject's current medication is changed as a result of study participation
* Outpatient >=12 years of age at Visit 1 who have had a diagnosis of asthma, as defined by the National Institutes of Health. Countries with local restrictions prohibiting enrolment of adolescents will only enroll subjects >=18 years of age
* Male or an eligible female. Eligible female is defined as having non-childbearing potential or having childbearing potential and using an acceptable method of birth control consistently and correctly.
* Best pre-bronchodilator FEV1 of 40% to 80% of their predicted normal value.
* Demonstrate >=12% and >=200 mL reversibility of FEV1 within 10 to 40 minutes following 4 inhalations of albuterol/salbutamol inhalation aerosol (or an equivalent nebulized treatment with albuterol/salbutamol solution) or have documented reversibility testing within the 6 months prior to Visit 1 meeting this measure of reversibility. A spacer device may be used for testing, if required.
* If subject have received ICS for at least 12 weeks prior to Visit 1 and their treatment during the 4 weeks immediately prior to Visit 1 consisted of either of the two regimens (a or b).a.) A stable mid-dose or high-dose of ICS alone (e.g., >=FP 250 mcg twice daily) or b.) A stable dose of a mid-dose ICS/LABA combination (e.g., FP/Salmeterol [SALM] 250/50 mcg twice daily) or an equivalent combination via separate inhalers.
* Use of ICS/LABA are not permitted with LABA on the day of Visit 1.
* Must be able to replace current SABA treatment with albuterol/salbutamol aerosol inhaler at Visit 1 for use as needed, during the study. Subjects must be able to withhold albuterol/salbutamol for at least 6 hours prior to study visits

Exclusion Criteria:

* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest or hypoxic seizures within the last 5 years.
* Upper or lower respiratory tract, sinus, or middle ear that is: not resolved within 4 weeks of Visit 1 and led to a change in asthma management or, in the opinion of the investigator, expected to affect the subject's asthma status or the subject's ability to participate in the study.
* Any asthma exacerbation that required oral corticosteroids within the 12 weeks prior to Visit 1 or, resulted in an overnight hospitalization requiring additional treatment for asthma within 6 months prior to Visit 1.
* A subject must not have current evidence of atelectasis (segmental or larger), bronchopulmonary dysplasia, chronic obstructive pulmonary disease, Or any evidence of concurrent respiratory disease other than asthma
* A subject must not have any clinically significant, uncontrolled condition or disease state that, in the opinion of the investigator, would put the safety of the subject at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study
* Chronic stable hepatitis B or C are acceptable provided their screening alanine transaminase (ALT) is <2x upper limit of normal (ULN) and the y otherwise meet the entry criteria. Chronic co-infection with both hepatitis B and hepatitis C are not eligible
* Clinical visual evidence of candidiasis at Visit 1
* Use of any investigational drug within 30 days prior to Visit 1 or within five half-lives (t½), whichever is longer of the two.
* Allergies to drug or milk protein: any adverse reaction, to any beta2-agonist, sympathomimetic drug, or any intranasal, inhaled, or systemic corticosteroid therapy or known or suspected sensitivity to the constituents of the NDPI, or history of severe milk protein allergy
* Administration of medication that would significantly affect the course of asthma, or interact with study drug
* Use of immunosuppressive medications during the study.
* Use of potent CYP3A4 inhibitor within 4 weeks of Visit 1.
* A subject or his/her parent or legal guardian has any infirmity, disability, disease, or resides in a geographical location which seems likely, in the opinion of the Investigator, to impair compliance with any aspect of this study protocol, including visit schedule, and completion of the daily diaries.
* Current smoker or has a smoking history of 10 pack-years (20 cigarettes/day for 10 years). A subject may not have used inhaled tobacco products within the past 3 months (i.e., cigarettes, cigars, or pipe tobacco).
* If subject is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.
* Subject previously randomized to treatment with FF/VI or FF in another Phase III study
* Subjects working on night shift a week prior to Visit 1 or during the study period.
* Adolescents who are wards of the state or government

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1040 (Actual)
Dates: Start 2012-09-20; Primary Completion 2013-10-01 (Actual); Study Completion 2013-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (112):
- United States (36):
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Rancho Mirage, California
  - GSK Investigational Site, Rolling Hills Estates, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Vista, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Wheat Ridge, Colorado
  - GSK Investigational Site, Tallahassee, Florida
  - GSK Investigational Site, Coeur d'Alene, Idaho
  - GSK Investigational Site, Normal, Illinois
  - GSK Investigational Site, Bethesda, Maryland
  - GSK Investigational Site, Columbia, Maryland
  - GSK Investigational Site, North Dartmouth, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Rolla, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Skillman, New Jersey
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Shelby, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Middleburg Heights, Ohio
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Fort Mill, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, El Paso, Texas
  - GSK Investigational Site, Waco, Texas
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Seattle, Washington
- Argentina (8):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Nueve de Julio, Buenos Aires
  - GSK Investigational Site, San Rafael, Mendoza Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Berazategui
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (7):
  - GSK Investigational Site, Rancagua, Reg Del Libert Bern Ohiggins
  - GSK Investigational Site, Quillota, Región de Valparaíso
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Germany (7):
  - GSK Investigational Site, Potsdam, Brandenburg
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Koblenz, Rhineland-Palatinate
  - GSK Investigational Site, Leipzg, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Großhansdorf, Schleswig-Holstein
  - GSK Investigational Site, Berlin
- Mexico (4):
  - GSK Investigational Site, Zapopan, Jalisco
  - GSK Investigational Site, Morelia, Michoacán
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
- Netherlands (7):
  - GSK Investigational Site, Almelo
  - GSK Investigational Site, Breda
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Enschede
  - GSK Investigational Site, Hoorn
  - GSK Investigational Site, Veldhoven
  - GSK Investigational Site, Zutphen
- Poland (6):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Tarnów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Romania (10):
  - GSK Investigational Site, Bacau
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Deva
  - GSK Investigational Site, Iași
  - GSK Investigational Site, Piteşti
  - GSK Investigational Site, Ploieşti
  - GSK Investigational Site, Timișoara
- Russia (15):
  - GSK Investigational Site, Blagoveshchensk
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Chita
  - GSK Investigational Site, Ivanovo
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Nizhny Novgorod
  - GSK Investigational Site, Pyatigorsk
  - GSK Investigational Site, Ryazan
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Stavropol
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Vladivostok
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yekaterinburg
- Sweden (5):
  - GSK Investigational Site, Gothenburg
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Luleå
  - GSK Investigational Site, Lund
  - GSK Investigational Site, Uppsala
- Ukraine (7):
  - GSK Investigational Site, Dnipropetrovsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kiev
  - GSK Investigational Site, Kyiv
  - GSK Investigational Site, Poltava
  - GSK Investigational Site, Vinnytsia
  - GSK Investigational Site, Zaporizhia

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- [Derived] Bernstein DI, Bateman ED, Woodcock A, Toler WT, Forth R, Jacques L, Nunn C, O'Byrne PM. Fluticasone furoate (FF)/vilanterol (100/25 mcg or 200/25 mcg) or FF (100 mcg) in persistent asthma. J Asthma. 2015;52(10):1073-83. doi: 10.3109/02770903.2015.1056350. Epub 2015 Aug 18. PMID 26291137
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 116863 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants meeting eligibility criteria at the Screening visit entered a 4-week Run-in Period for Baseline safety evaluations and measures of asthma status. Participants were then randomized to a 12-week Treatment Period. A total of 2019 participants were screened; 1039 were randomized and received >=1 dose of study treatment.
Pre-assignment Details: One participant was determined to have been randomized at each of two United States sites. Upon discovery of the duplicate enrollment, the participant was withdrawn. To account for only one randomization by this participant, a total randomized population of 1039 was used as the basis for the study analysis.
Groups:
- FF 100 µg OD: Participants received Fluticasone Furoate (FF) 100 microgram (µg) inhalation powder once daily (OD) in the evening from a dry powder inhaler (DPI) for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FF/VI 100/25 µg OD: Participants received FF/Vilanterol (VI) 100/25 µg inhalation powder OD in the evening from a DPI for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FF/VI 200/25 µg OD: Participants received FF/VI 200/25 µg inhalation powder OD in the evening from a DPI for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
Period: Overall Study
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Started | 347 | 346 | 346
Completed | 296 | 314 | 321
Not Completed | 51 | 32 | 25
Not completed — Lack of Efficacy | 33 | 13 | 11
Not completed — Withdrawal by Subject | 8 | 8 | 5
Not completed — Physician Decision | 3 | 4 | 4
Not completed — Adverse Event | 4 | 3 | 3
Not completed — Protocol Violation | 2 | 3 | 0
Not completed — Protocol-defined Stopping Criteria | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- FF 100 µg OD: Participants received FF 100 µg inhalation powder OD in the evening from a DPI for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- FF/VI 100/25 µg OD: Participants received FF/VI 100/25 µg inhalation powder OD in the evening from a DPI for 12 weeks. Participants were provided albuterol/salbutamol inhalation aerosol to be used as rescue medication during the Treatment Period.
- Total: Total of all reporting groups
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD | Total
Number analyzed (Participants) | 347 | 346 | 346 | 1039
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.7 (15.89) | 45.9 (16.14) | 46.6 (14.72) | 45.7 (15.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 199 | 205 | 224 | 628
  Male | 148 | 141 | 122 | 411
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 26 | 20 | 28 | 74
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian - East Asian Heritage | 0 | 1 | 0 | 1
  Asian - Japanese Heritage | 1 | 0 | 0 | 1
  Asian - South East Asian Heritage | 3 | 1 | 2 | 6
  Native Hawaiian or other Pacific Islander | 0 | 1 | 0 | 1
  White - White/Caucasian/European Heritage | 305 | 307 | 300 | 912
  Mixed Race | 12 | 16 | 13 | 41
  Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weighted Mean Forced Expiratory Volume in One Second (FEV1) Over 0 to 24 Hours Post-dose at the End of the 12-week Treatment Period
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. The weighted mean was calculated from the pre-dose FEV1 (within 30 minutes prior to dosing) and post-dose FEV1 measurements at 5, 15, and 30 minutes and at 1, 2, 3, 4, 5, 12, 16, 20, 23, and 24 hours on Day 84/Week 12. At each time point, the highest of three technically acceptable measurements was recorded. Change from Baseline was calculated as the weighted mean of the 24-hour serial FEV1 measures on Day 84/Week 12 minus the Baseline value. Baseline was the pre-dose FEV1 measurement value obtained at Visit 3. The analysis was performed using an Analysis of Covariance (ANCOVA) model with covariates of Baseline FEV1, region, sex, age, and treatment.
Time Frame: Baseline and Week 12
Population: Intent-to-Treat (ITT) Population: all participants randomized to treatment, who received at least one dose of the study medication. Only those participants with non-missing covariates and Week 12 weighted mean data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 288 | 312 | 312
Liters | 0.366 (0.0231) | 0.474 (0.0221) | 0.499 (0.0222)
Statistical Analysis 1: Comparison: FF 100 µg OD vs FF/VI 100/25 µg OD; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = 0.108, 95% CI 2-sided [0.045 to 0.171]
Statistical Analysis 2: Comparison: FF/VI 100/25 µg OD vs FF/VI 200/25 µg OD; Test type: Superiority or Other; Mean Difference (Final Values) = 0.024, 95% CI 2-sided [-0.037 to 0.086]

2. Secondary Outcome: Change From Baseline in Clinic Visit Trough FEV1 at the End of the 12-week Treatment Period
Description: Pulmonary function was measured by FEV1, defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 is defined as a pre-dose FEV1 measurement taken at a clinic visit while still on-treatment. Change from Baseline in trough FEV1 at the end of the 12-week treatment period was defined using the 24-hour post-dose serial FEV1 measurement taken at the Week 12 clinic visit. Change from Baseline was calculated as the Week 12 trough FEV1 value minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline trough FEV1, region, sex, age, and treatment. The last observation carried forward (LOCF) method was used to impute missing data, in which the last non-missing post-Baseline on-treatment measurement at scheduled clinic visits was used to impute the missing measurements.
Time Frame: Baseline and Week 12
Population: ITT Population. Only those participants with non-missing covariates and post-Baseline FEV1 data were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 336 | 334 | 337
Liters | 0.365 (0.0220) | 0.441 (0.0221) | 0.457 (0.0220)

3. Secondary Outcome: Change From Baseline in the Percentage of Rescue-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: The number of inhalations of rescue albuterol/salbutamol inhalation aerosol used during the day and night was recorded by the participants in a daily electronic diary (eDiary). A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no use of rescue medication was considered to be rescue free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 12-week treatment period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of rescue-free 24-hr periods
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 346 | 345 | 346
Percentage of rescue-free 24-hr periods | 22.6 (1.84) | 34.8 (1.85) | 35.8 (1.85)

4. Secondary Outcome: Change From Baseline in the Percentage of Symptom-free 24-hour (hr) Periods During the 12-week Treatment Period
Description: Asthma symptoms were recorded in a daily eDairy by the participants every day in the morning and evening before taking any rescue or study medication and before the peak expiratory flow measurement. A 24-hour (hr) period in which a participant's responses to both the morning and evening assessments indicated no symptoms was considered to be symptom free. The Baseline value was derived from the last 7 days of the daily eDiary prior to the randomization of the participant. Change from Baseline was calculated as the averaged value during the 12-week treatment period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Percentage of symptom-free 24-hr periods
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 346 | 345 | 346
Percentage of symptom-free 24-hr periods | 19.4 (1.74) | 27.2 (1.74) | 29.0 (1.74)

5. Secondary Outcome: Change From Baseline in Daily Morning (AM) Peak Expiratory Flow (PEF) Averaged Over the 12-week Treatment Period
Description: Peak Expiratory Flow (PEF) is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use and each morning. The best of three measurements was recorded. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily AM PEF over the 12-week treatment period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 346 | 345 | 345
Liters per minute | 19.1 (2.25) | 44.3 (2.25) | 47.7 (2.25)

6. Secondary Outcome: Change From Baseline in Daily Evening (PM) PEF Averaged Over the 12-week Treatment Period
Description: PEF is defined as the maximum airflow during a forced expiration beginning with the lungs fully inflated. PEF was measured by the participants using a hand-held electronic peak flow meter each evening prior to the dose of study medication and any rescue albuterol/salbutamol inhalation aerosol use and each morning. The best of three measurements was recorded. Change from Baseline (defined as the last 7 days prior to randomization of the participants) was calculated as the value of the averaged daily PM PEF over the 12-week treatment period minus the Baseline value. The analysis was performed using an ANCOVA model with covariates of Baseline, region, sex, age, and treatment.
Time Frame: Baseline and Weeks 1-12
Population: ITT Population. Only those participants available at the specified time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Liters per minute
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Number analyzed (Participants) | 346 | 345 | 346
Liters per minute | 15.5 (2.24) | 39.7 (2.24) | 41.7 (2.24)

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) and non-serious AEs were collected from the first dose of study medication up to Week 12/Early Withdrawal.
Description: SAEs and AEs were collected in members of Intent-to-Treat (ITT) Population, comprised of all participants randomized to treatment who received at least one dose of the study medication.
Arm/Group | FF 100 µg OD | FF/VI 100/25 µg OD | FF/VI 200/25 µg OD
Serious Adverse Events (participants affected / at risk) | 3/347 | 4/346 | 1/346
Other Adverse Events (participants affected / at risk) | 67/347 | 54/346 | 52/346
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg OD (N=347) | FF/VI 100/25 µg OD (N=346) | FF/VI 200/25 µg OD (N=346)
Pneumonia (Infections and infestations) | 2 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Borderline mucinous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 1 | 0
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 µg OD (N=347) | FF/VI 100/25 µg OD (N=346) | FF/VI 200/25 µg OD (N=346)
Nasopharyngitis (Infections and infestations) | 26 | 22 | 25
Upper respiratory tract infection (Infections and infestations) | 12 | 8 | 7
Headache (Nervous system disorders) | 32 | 29 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.